CLINICAL TRIAL: NCT02633735
Title: EHR-based Decision Support for Pediatric Acute Abdominal Pain in Emergency Care
Acronym: Appy-CDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Kaiser Permanente (Other); Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-025
Record Dates: First submitted 2015-11-24; First posted 2015-12-17 (Estimated); Results first posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2019-09

CONDITIONS: Appendicitis
Keywords: Clinical Decision Support
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Intervention Model Description: Parallel cluster-randomized clinical trial at 14 general EDs in two large care system to evaluate the impact of appy-CDS intervention with a pre and post intervention phases
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Appy CDS (Experimental): The Appy-cds intervention is a point of care clinical decision support system designed to identify pediatric patients at risk for appendicitis using EHR and supplemental data. The intervention is administered to providers in this arm.
  Interventions: Other: Appy CDS
- Usual Care (No Intervention)

INTERVENTIONS:
Other: Appy CDS — See description under arm/group section
  Arms: Appy CDS

SUMMARY:
Although appendicitis is the most common surgical emergency in children, its diagnosis remains a challenge and thus, emergency department (ED) providers increasingly rely on computed tomography to distinguish appendicitis from other conditions. This project (a) uses electronic health record (EHR) technology to deliver patient-specific clinical decision support to ED providers at the point of care, (b) assesses the impact of this intervention on the use of diagnostic imaging and clinical outcomes, and (c) assesses the impact of the intervention on the costs of care delivered. This innovative project will be a template for extending EHR-based clinical decision support to other domains of emergency care to ultimately improve a broad range of pediatric acute care outcomes.

The proposed intervention, referred to as appy-CDS, is specifically designed for widespread use in EDs and could reduce reliance on advanced diagnostic imaging for pediatric and adolescent patients with acute abdominal pain while maintaining or improving clinical outcomes. Investigators aim to develop and implement an interactive, evidence-based clinical decision support tool to optimize care for children and adolescents presenting to a general or non-pediatric ED with acute abdominal pain.

DETAILED DESCRIPTION:
Abdominal pain is one of the most common reasons for children and adolescents to seek care in the emergency department (ED). Computed tomography (CT) has been promoted as a method to improve diagnostic accuracy when evaluating patients with acute abdominal pain. In the past 20 years, CT use has increased dramatically, especially for children receiving care in general ED settings. Although in some adult cohorts, increased CT use has been associated with decreased rates of negative appendectomies, similar improvements in health outcomes among children with acute abdominal pain have not occurred. Negative consequences of CT include increased costs and substantial exposure to ionizing radiation.

Although appendicitis is the most common surgical emergency in children, its diagnosis remains a challenge and thus, emergency department (ED) providers increasingly rely on computed tomography to distinguish appendicitis from other conditions. This project (a) uses electronic health record (EHR) technology to deliver patient-specific clinical decision support to ED providers at the point of care, (b) assesses the impact of this intervention on the use of diagnostic imaging and clinical outcomes, and (c) assesses the impact of the intervention on the costs of care delivered.

The proposed intervention, referred to as appy-CDS, is specifically designed for widespread use in EDs and could reduce reliance on advanced diagnostic imaging for pediatric and adolescent patients with acute abdominal pain while maintaining or improving clinical outcomes. This cluster randomized trial builds on more than 10 years of work on derivation and validation of ED-based clinical decision rules, previous successful outpatient and emergency department clinical decision support interventions, and complex economic and statistical analyses of risk assessment and ED resource use. In this project, the investigators aim to extend the benefits of previous efforts by developing and implementing an interactive, evidence-based clinical decision support tool to optimize care for children and adolescents presenting to a general or non-pediatric ED with acute abdominal pain. The results of this project will extend the understanding of how to maximize the clinical return on massive public and private sector investments being made in sophisticated EHR systems. If successful, this flexible decision support tool could be adapted and implemented broadly in a range of acute care settings to both standardize and personalize care delivered to pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents ages 5-20 years with abdominal pain
* internal med, family med, or emergency med trained providers at participating EDs

Exclusion Criteria:

* select comorbid conditions
* previous abdominal surgery
* treated for select comorbid conditions

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5940 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elyse O Kharbanda, MD, MPH, Principal Investigator — HealthPartners Institute; Anupam B Kharbanda, MD, MSc, Principal Investigator — Children's Hospital and Clinics of Minnesota
Locations (2):
- United States (2):
  - Kaiser Permanente Northern California, Oakland, California
  - HealthPartners Medical Group, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kharbanda AB, Vazquez-Benitez G, Ballard DW, Vinson DR, Chettipally UK, Dehmer SP, Ekstrom H, Rauchwerger AS, McMichael B, Cotton DM, Kene MV, Simon LE, Zhu J, Warton EM, O'Connor PJ, Kharbanda EO; Clinical Research on Emergency Services and Treatments Network (CREST) and the Critical Care Research Center, HealthPartners Institute. Effect of Clinical Decision Support on Diagnostic Imaging for Pediatric Appendicitis: A Cluster Randomized Trial. JAMA Netw Open. 2021 Feb 1;4(2):e2036344. doi: 10.1001/jamanetworkopen.2020.36344. PMID 33560426
- [Derived] Cotton DM, Vinson DR, Vazquez-Benitez G, Margaret Warton E, Reed ME, Chettipally UK, Kene MV, Lin JS, Mark DG, Sax DR, McLachlan ID, Rauchwerger AS, Simon LE, Kharbanda AB, Kharbanda EO, Ballard DW; Clinical Research on Emergency Services and Treatments (CREST) Network. Validation of the Pediatric Appendicitis Risk Calculator (pARC) in a Community Emergency Department Setting. Ann Emerg Med. 2019 Oct;74(4):471-480. doi: 10.1016/j.annemergmed.2019.04.023. Epub 2019 Jun 19. PMID 31229394

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: ED Sites were randomized to the AppyCDS intervention or usual care (UC). Sites were stratified by health system and then grouped on patterns of pediatric referral and provider cross coverage. EDs or groups of EDs were sorted into pairs by estimated pediatric patient volume. Study phases were consistent but date ranges varied by health system.
Groups:
- Control: Usual care
- Intervention: The appy-cds intervention is a point of care clinical decision support system designed to identify pediatric patients at risk for appendicitis using EHR and supplemental data. The appy-cds has multiple components, 1) presents risk prediction/stratification to provider, 2) provides recommendations consistent with standardized appendicitis care, 3) alerts for unnecessary exposure to ionizing radiation via a best practice alert. The intervention is administered to providers in this arm.
  appy-cds: See description under arm/group section
Period: Pre-implementation Phase
Arm/Group | Control | Intervention
Started | 788 | 1011
Completed | 788 | 1011
Not Completed | 0 | 0
Period: Implementation Phase
Arm/Group | Control | Intervention
Started | 1991 | 2150
Completed | 1991 | 2150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline characteristics reflect the sum of participants who completed the pre-implementation and implementation phase in both study arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 2779 | 3161 | 5940
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.7 (4.5) | 11.9 (4.6) | 11.8 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1512 | 1780 | 3292
  Male | 1267 | 1381 | 2648
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 788 | 1104 | 1892
  Not Hispanic or Latino | 1991 | 2057 | 4048
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 176 | 367 | 543
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 402 | 473 | 875
  White | 2000 | 2059 | 4059
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 201 | 262 | 463

OUTCOME MEASURES:

1. Primary Outcome: Pre to Post Ratio of Image Use
Description: First, we evaluated whether patient characteristics (age, sex, race/ethnicity) differed by study arm and phase using frequency distributions, means and standard deviations. Second, we estimated use of imaging for CT, US and CT or US by study arm and phase. We evaluated the effectiveness of AppyCDS by estimating the ratio of ratios (ROR) and 95% confidence intervals (CI) of intervention arm, from pre-intervention phase to intervention phase as compared to UC arm over the two study phases, for all imaging outcomes.
Time Frame: pre-intervention of 8 months (average), and post intervention of 23 months
Population: Numbers are sum of subjects in pre-implementation and implementation phases.
Measure: Mean (95% Confidence Interval); unit: ratio of pre-post use
Arm/Group | Control | Intervention
Number analyzed (Participants) | 2779 | 3161
ratio of pre-post use
  CT Use | 1.13 [.92 to 1.4] | 1.07 [.97 to 1.17]
  US Use | 1.03 [.92 to 1.16] | 1.01 [.91 to 1.12]
  All Imaging Use | 1.06 [.98 to 1.14] | 1.02 [.94 to 1.11]

ADVERSE EVENTS:
Time Frame: Within 7 days of index ED visit.
Description: The number analyzed are the sum of participants who completed the pre-implementation and implementation phase in both study arms. Negative appendicitis and appendiceal perforation were monitored for the subset of participants that had a surgical procedure following exposure to the clinical decision support intervention.
Groups:
- Appy CDS Intervention: The Appy-cds intervention is a point of care clinical decision support system designed to identify pediatric patients at risk for appendicitis using EHR and supplemental data. The Appy-cds has multiple components, 1) presents risk prediction/stratification to provider, 2) provides recommendations consistent with standardized appendicitis care, 3) alerts for unnecessary exposure to ionizing radiation via a best practice alert. The intervention is administered to providers in this arm.
  Post Appy Clinical Decision Support: The Appy CDS is a point of care clinical decision support system that provides the provider with 1) risk for appendicitis based on EHR data, 2) recommendations on actions to take based on risk, 3) advises on imaging use.
- Control: People in the control arm receive usual care.
Arm/Group | Appy CDS Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/3161 | 0/2779
Serious Adverse Events (participants affected / at risk) | 96/3161 | 109/2779
Other Adverse Events (participants affected / at risk) | 222/3161 | 224/2779
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Appy CDS Intervention (N=3161) | Control (N=2779)
Appendiceal perforation (Gastrointestinal disorders) | 63/402 | 67/341
Negative appendicitis (Surgical and medical procedures) | 20/421 | 27/365
Missed appendicitis (General disorders) | 13 | 15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Appy CDS Intervention (N=3161) | Control (N=2779)
Return to ED within 7 days of index (General disorders) | 222 | 224

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/35/NCT02633735/Prot_SAP_000.pdf